CLINICAL TRIAL: NCT03822559
Title: A Randomized, Double-masked, Controlled Parallel Group, Multi-center Study of DE-111A (Fixed Dose Combination of Tafluprost and Timolol Eye Drops) on the Treatment of Open Angle Glaucoma or Ocular Hypertension (With Tafluprost Eye Drops as a Comparator)
Brief Title: A Study of DE-111A on the Treatment of Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0111A04LT
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Open-angle Glaucoma, Ocular Hypertension
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — tafluprost; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DE-111A eye drops (Experimental)
  Interventions: Drug: A preservative-free, a clear, colorless sterile aqueous ophthalmic solution containing 0.015mg of tafluprost and 5.0mg of timolol in 1mL
- 0.0015% tafluprost eye drops (Active Comparator)
  Interventions: Drug: A preservative-free, a clear, colorless sterile aqueous ophthalmic solution containing 0.015mg of tafluprost in 1mL

INTERVENTIONS:
Drug: A preservative-free, a clear, colorless sterile aqueous ophthalmic solution containing 0.015mg of tafluprost and 5.0mg of timolol in 1mL — One drop a time, once daily administration of DE-111A eye drops in the affected eye(s) at 8:00 am (±1h) for 3 months.
  Arms: DE-111A eye drops
Drug: A preservative-free, a clear, colorless sterile aqueous ophthalmic solution containing 0.015mg of tafluprost in 1mL — One drop a time, once daily administration of preservative-free 0.0015% tafluprost eye drops in the affected eye(s) at 8:00 (±1h) for 3 months.
  Arms: 0.0015% tafluprost eye drops

SUMMARY:
The objective of this study is to investigate whether the IOP (intraocular pressure) -lowering effect of DE-111A (preservative-free fixed dose combination of 0.0015% tafluprost and 0.5% timolol eye drops, administered one drop a time, once daily for 3 months) is superior to the monotherapy of tafluprost 0.0015% eye drops administered one drop a time, once daily for 3 months) in subjects with open-angle glaucoma or ocular hypertension in China as well as comparison of safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma (including primary open angle glaucoma, exfoliation glaucoma or pigmentary glaucoma) in one or both eyes or ocular hypertension for which the subject has been using prostaglandin or beta-adrenergic blocker IOP (intraocular pressure) -lowering drugs before the screening visit
* Those who have signed the informed consent form

Exclusion Criteria:

* Women who are pregnant, nursing or planning pregnancy, or women of child-bearing potential who are not using a reliable method of contraception
* Anterior chamber angle in either eye to be treated with the level <2 according to Shaffer classification as measured by gonioscopy
* Corneal disorder or other disease preventing reliable applanation tonometry in the treated eyes, including refractive surgery of ocular anterior segment)
* Alcohol or drug abuse
* Current participation in another clinical trial involving an investigational drug/device, or participation in such a trial within 30 days before Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average diurnal IOP (intraocular pressure) | Three months
  Diurnal IOP measurements will be performed at 8:00 (±1 h), 10:00 (±1 h) and 16:00 (±1 h).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Aier Eye Hospital Group Co., Ltd Changsha Aier Eye Hospital, Changsha
  - Eye & Ent Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No